CLINICAL TRIAL: NCT06677021
Title: Evaluation of Physical Activity Behaviours, and Psychosocial Health Outcomes in Children and Young People with Chronic Kidney Disease
Brief Title: Understanding Physical Activity and Quality of Life in Children and Young People with Chronic Kidney Disease
Acronym: PA-QOL-CKD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Margaret University (Other)
Responsible Party: Principal Investigator, Pelagia Koufaki, PhD, Reader in Exercise Physiology and Rehabilitation Sciences, Queen Margaret University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: BUR 23-23
Record Dates: First submitted 2024-11-01; First posted 2024-11-06 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Chronic Kidney Disease Stages 3-5
Keywords: Children and Young People; Chronic Kidney Disease; Physical activity; Psychosocial outcomes; Quality of life; Adolescents; Children; Exercise; Mental Health
MeSH Terms: conditions — Renal Insufficiency, Chronic; Motor Activity; Psychological Well-Being | interventions — Exercise; Quality of Life

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Physcial Activity Exercises (Other)
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — Physical activity promotion and engagement
  Other Names: Quality of life

SUMMARY:
Children and young people (CYP) with chronic kidney disease (CKD) say that physical activity, school, social activities and tiredness are the main issues they want to improve. As CKD in CYP is a rare disease, there is not much research into understanding these aspects, making it difficult to know how to support patients better. This project aims to investigate how physically active CYP with CKD are, and what psychosocial factors are affected by their illness. CYP aged 6-18 will take part in a battery of physical activity tests, par-take in an online survey looking at physical activity, quality of life, mental health, fatigue and strengths and difficulties, and take part in an interview to better understand what it is like to live with CKD.

DETAILED DESCRIPTION:
The aim of this research is to document and evaluate the relationship between physical activity patterns and behaviours and psychosocial outcomes in children and young people with CKD. A second aim is to explore through qualitative methods contextual factors that may explain the type, direction and nature of relationships identified in the quantitative phase.

This research will be conducted in multiple phases to maximise recruitment.

1. Phase 1 consists of a battery of in-person physical functioning tests.
2. Phase 2 consists of an online survey of validated questionnaires.
3. Phase 3 consists of online or in-person interviews with CYP

Participants recruited through NHS Scotland will take part in all 3 phases. Only Phase 2 (online survey) will additionally be disseminated through patient organisations across the UK to maximise recruitment.

In phase 1, participants will take part in a battery of physical activity functioning assessments including multistage bleep tests, sit-up tests, and handgrip tests. Participants will also be given an accelerometer measure to track movements over 7 days. Participants taking part in this phase will also complete the phase 2 online survey which includes a physical activity, Quality of life, Fatigue, Strength and Difficulties, and Mental health questionnaire.

In phase 3, participants from phase 1 will return and take part in an interview to gain deeper insights into psychosocial influences and limitations in engaging in physical activity as well as gaining a better understanding of the impact of CKD on psychosocial wellbeing.

ELIGIBILITY:
Inclusion Criteria:

* CYP of school age between 6 and 18 years
* Living and receiving care in Scotland for CKD
* no clinical contradictions to physical function assessments

Exclusion Criteria:

* Enrolment in other clinical trials in which treatment is masked/blinded
* Deemed to be clinically unstable by treating physician for participating in physical activity and exercise
* Severe cognitive impairment (as will be unable to give consent)
* Aged <6 or >18 years.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Physical Activity: cardiorespiratory fitness | Baseline
  Multistage Bleep Test - This test entails a progressively incremental jogging/running challenge along a 20-meter distance while keeping to an auditory signal. The test is terminated when participants cannot maintain pace to the auditory signal or upon participant refusal to continue.
Physical Activity: forearm strength | Baseline
  Handgrip test - This test assesses static forearm strength using a handheld dynamometer.
Physical Activity: muscular endurance | Baseline
  Sit-up test - This test will assess muscular endurance, particularly abdominal strength (dynamic trunk strength).
Accelerometer | Baseline
  Participants will be given an accelerometer to be worn around their wrist. This device tracks step counts continuously for 7-days. Average daily step counts, and average sedentary time will be calculated.

SECONDARY OUTCOMES:
Frequency of physical activity | Baseline
  The Physical Activity Questionnaire for older children (PAQ-C) aged 8-14 will be used to measure general levels of PA throughout the school year.
  Physical activity summary score will be calculated on a scale from 1-5. A score of 1 indicates low physical activity, whereas a score of 5 indicates high physical activity.
Frequency of physical activity | Baseline
  The Physical Activity Questionnaire for adolescents (PAQ-A) aged 14-18 will be used to measure general levels of PA throughout the school year.
  Physical activity summary score will be calculated on a scale from 1-5. A score of 1 indicates low physical activity, whereas a score of 5 indicates high physical activity.
Quality of Life | Baseline
  The multidimensional Paediatric Quality of Life Inventory (PedsQLv4) questionnaire will be used to estimate scores that reflect the domains of physical functioning, emotional functioning, social functioning, and school functioning.
  A quality of life score will be calculated on a scale from 0-100. Higher scores = Better HRQOL.
Fatigue | Baseline
  The multidimensional Fatigue scale (PedsQLv3 Fatigue) questionnaire will be used to estimate scores that reflect the domains of general fatigue, sleep/rest fatigue and cognitive fatigue.
  A Fatigue HRQOL score will be calculated on a scale from 0-100. Higher scores = Better HRQOL and fewer problems or symptoms
Mental Health | Baseline
  The Revised Child Anxiety and Depression Scale (RCADS) will be used to estimate scores related to the following subscales: separation anxiety disorder, social phobia, generalized anxiety disorder, panic disorder, obsessive compulsive disorder, and low mood (major depressive disorder).
  Each subscale will be calculated on a scale ranging from 0-18 and 0-30. From this t-scores can be calculated.
  Low severity: T-score below 65 Medium severity: T-score between 65-70 High severity: T-score above 70
Strengths and Difficulties | Baseline
  The Strength and Difficulties Questionnaire (SDQ) will be used to estimate scores related to the following subscales: emotional symptoms, conduct problems, hyperactivity/inattention, peer relationship problems, prosocial behaviour.
  A Total difficulties score will be calculated on a scale from 0-40. Higher scores = more difficulties.
Qualitative exploration of experiences, attitudes, and preferences | within 1-2months after primary outcomes have been completed
  Semi structured interviews with participants and families will be used to to gain deeper insights into patient experiences, attitudes, preferences, and future direction

CONTACTS AND LOCATIONS:
Locations (1):
- Glasgow Royal Hospital for Children, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No Plan yet